CLINICAL TRIAL: NCT00083928
Title: A Phase 2 Randomized, Double-Blind Trial of the Clinical Activity and Safety of Å6 in Patients With Asymptomatic CA125 Progression of Epithelial Ovarian Cancer After First-Line Chemotherapy
Brief Title: Efficacy of Å6 in Ovarian Cancer Patients Following First-Line Chemotherapy and a Rising CA125 Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ångstrom Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Å6-003
Record Dates: First submitted 2004-06-03; First posted 2004-06-07 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Ovarian Cancer; Primary Peritoneal Carcinoma
Keywords: Asymptomatic; subcutaneous; CA125 Progression; Angstrom; Ångstrom; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

INTERVENTIONS:
Drug: Å6 subcutaneous injection

SUMMARY:
The purpose of this study is to determine whether injections of Å6 are effective in treating ovarian cancer patients who have completed first-line therapy and currently have no detectable cancer but have experienced a doubling of CA 125 levels.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥18 years of age
* Histologically or cytologically documented primary epithelial ovarian carcinoma, cancer of the Fallopian tube, or primary peritoneal carcinoma
* Completion of first-line chemotherapy
* Clinical remission as a result of chemotherapy
* History of normal CA125 level after initial course of therapy
* CA125 serum level has shown 2 consecutive rises based on 3 consecutive samples which are mutually >= 28 days apart, provided that:

  1. the 3rd sample is above the institution's ULN, and
  2. the 3rd sample is confirmed by a 4th sample which is likewise higher than the 2nd sample value and is above the institution's ULN
* No clinically evident disease progression, as assessed by history, physical examination, computed tomographic (CT) scan, or magnetic resonance imaging (MRI)
* ECOG Performance Status of 0 or 1
* No clinically significantly abnormal clinical laboratory tests or concomitant illnesses
* Ability and willingness to self-administer subcutaneous injections
* Although pregnancy is extremely unlikely in this patient population because of the disease and prior treatment, patients who have the potential to become pregnant must have a negative pregnancy test and must agree to practice an effective method of contraception throughout the trial.

Exclusion Criteria:

* Persistent adverse events due to agents administered more than 4 weeks earlier
* More than 1 course of previous chemotherapy for the qualifying cancer
* Disease requiring chemotherapy or radiotherapy
* Ascites
* Recent history of active infection, gastrointestinal bleeding, thromboembolic disorders, or anticoagulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-02 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - California Oncology of the Central Valley, Fresno, California
  - USC Keck School of Medicine Women's and Childrens Hospital, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - UC Davis Health System, Sacramento, California
  - Scripps Cancer Center, San Diego, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Medical College of Georgia Dept. of OB/GYN, Saint Agusta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Gynecologic Oncology, Hinsdale, Illinois
  - St. Vincent Gyn-Onc, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Louisville JG Brown Cancer Center, Louisville, Kentucky
  - Hematology & Oncology Specialists, New Orleans, Louisiana
  - Barnes Jewish Hospital, St Louis, Missouri
  - Gabrail Cancer Center, Canton, Ohio
  - OSU College of Medicine, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Gynecologic-Oncology Research and Development, LLC, Greenville, South Carolina
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia